CLINICAL TRIAL: NCT03712436
Title: A Study of Early Palliative Care in Newly Diagnosed Cancer Patients at Black Lion Hospital, Addis Ababa, Ethiopia
Brief Title: Examining Early Palliative Care in Newly Diagnosed Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2000023057
Record Dates: First submitted 2018-09-14; First posted 2018-10-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cancer
Keywords: Palliative Care; Supportive Care; Low Income Setting; LMIC; Africa
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of standard oncologic care versus standard oncologic care plus palliative care in a newly diagnosed oncology population.
Who Masked: Participant, Care Provider
Masking Description: blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving palliative care (Experimental): Patients receiving standard oncologic care plus palliative care.
  Interventions: Combination Product: Palliative care
- patients receiving standard oncological care (Active Comparator): Patients receiving standard oncologic care.
  Interventions: Combination Product: Standard oncological care

INTERVENTIONS:
Combination Product: Palliative care — The Palliative Care Package is a protocol for Palliative Care delivery, derived from the African Palliative Care Association and adapted to the local environment in Addis Ababa.
  Arms: patients receiving palliative care
Combination Product: Standard oncological care — Standard Oncological Care available in Addis Ababa, Ethiopia which includes chemotherapy, radiation oncology
  Arms: patients receiving standard oncological care

SUMMARY:
To understand the impact of initiation of palliative care in this low-resource setting, and whether palliative care is a cost-reducing intervention that will improve patient-reported outcomes and quality of life.

DETAILED DESCRIPTION:
The investigators overall goal is to understand the impact of initiation of early palliative care in an oncology population in a low-resource setting in order to provide guidance for future public health policies surrounding the provision of palliative care in Ethiopia. Hypothesis: The investigators hypothesize that initiation of palliative care in this low-resource setting is a cost-reducing intervention that will improve patient-reported outcomes and quality of life. Preliminary data: This research will focus on adult patients with oncologic diagnoses as preliminary research in this setting revealed that this patient population had the highest depression and anxiety scores, the lowest palliative outcome scores, and reported the highest costs of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any newly diagnosed cancer who are ambulatory and able to respond verbally to questions, are eligible for inclusion.

Exclusion Criteria:

* Patients who have not been diagnosed with cancer.
* Patients with diagnoses made more than 4 weeks ago, who are non-ambulatory, or are already receiving palliative care, are ineligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
African Palliative Care Association Palliative Outcome Scale (APCA POS) score | upon enrollment
  APCA POS: APCA POS measures unpleasant symptoms (pain, worry, other symptoms) on a scale of 0-5 (best to worst). We will measure at baseline.
African Palliative Care Association Palliative Outcome Scale (APCA POS) score | 12 weeks
  APCA POS: APCA POS measures unpleasant symptoms (pain, worry, other symptoms) on a scale of 0-5 (best to worst). We will compare baseline score to follow up score. An APCA POS score decrease of 3 from baseline will be signficant.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Score (HADS) | upon enrollment
  HADS score measures anxiety and depression on a scale of 0-3 (best to worst). We will measure at baseline.
Hospital Anxiety and Depression Score (HADS) | 12 weeks
  HADS score measures anxiety and depression on a scale of 0-3 (best to worst). HADS score decrease from baseline, as measured at follow up.

OTHER OUTCOMES:
Healthcare Usage | upon enrollment
  Evaluating the direct costs of all medical care,
Healthcare Usage | 8 weeks
  Evaluating the direct costs of all medical care.
Patient reported costs | 12 weeks
  Change in patient reported costs

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Reid, MD, Principal Investigator — Yale University
Locations (1):
- Black Lion Hospital Oncology Clinic, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reid E, Abathun E, Diribi J, Mamo Y, Hall P, Fallon M, Wondemagegnhu T, Grant L. Rationale and study design: A randomized controlled trial of early palliative care in newly diagnosed cancer patients in Addis Ababa, Ethiopia. Contemp Clin Trials Commun. 2020 Apr 6;18:100564. doi: 10.1016/j.conctc.2020.100564. eCollection 2020 Jun. PMID 32309673
- See also: HADS — http://www.svri.org/sites/default/files/attachments/2016-01-13/HADS.pdf
- See also: APCA POS — https://pos-pal.org/maix/apca-african-pos.php